CLINICAL TRIAL: NCT02777736
Title: Study Evaluating Relapses in Central Nervous System in Patients With Diffuse Large B-Cell Lymphoma Treated With Chemotherapy With or Without CNS Prophylaxis. Multicentric, Prospective, Randomized Phase III Study
Brief Title: CNS Prophylaxis in Diffuse Large B-cell Lymphoma
Acronym: CLSG-CNS-001
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Czech Lymphoma Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLSG-CNS-001; 2015-000591-97 (EudraCT Number)
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma, B cell; Central nervous system relapse; Methotrexate; Intrathecal chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A - Methotrexate i.v. (Experimental): Patients with risk factors for CNS relapse ≥ 2 or with occult meningeal involvement will receive 2 cycles of methotrexate 3g/m2 i.v. after the 3rd and 6th cycle of systemic chemotherapy (R CHOP or DA EPOCH R).
  Interventions: Drug: Methotrexate
- Arm B - Methotrexate i.t. (Active Comparator): Patients with risk factors for CNS relapse ≥ 2 or with occult meningeal involvement will receive intrathecal methotrexate 12mg in each cycle of systemic chemotherapy (6x).
  Interventions: Drug: Methotrexate
- Arm C - no Methotrexate (No Intervention): Patients with 0-1 risk factor for CNS relapse will not receive CNS prophylaxis.

INTERVENTIONS:
Drug: Methotrexate — i.v. or intrathecal CNS prophylaxis
  Other Names: Methotrexate,manufactured by EBEWE; Methotrexate, manufactured by HOSPIRA
  Arms: Arm A - Methotrexate i.v.; Arm B - Methotrexate i.t.

SUMMARY:
Comparison of cumulative incidence of CNS relapses in patients with diffuse large B-cell lymphoma with intermediate or high risk of CNS relapse treated with CNS prophylaxis: either with 2 doses of intravenous methotrexate 3g/m2 i.v.(arm A) or 6 doses of intrathecal methotrexate 12mg (arm B) and in patients with low risk of CNS relapse without CNS prophylaxis (arm C).

DETAILED DESCRIPTION:
Patients with diffuse large B-cell lymphoma are evaluated for risk factors of CNS relapse during initial staging (age > 60years, lactate dehydrogenase (LDH) > reference range, clinical stage III/IV, performance status according to Eastern Cooperative Oncology Group (ECOG) >1, kidney and/or adrenal gland involvement, involvement > 1 extranodal organ) including evaluation of cerebrospinal fluid.

All patients with systemic DLBCL without CNS involvement are treated with systemic chemotherapy: either 6 cycles of R CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednison) +2xR (rituximab) or 6 cycles of DA EPOCH R (dose adjusted etoposide, prednison, vincristin, cyclophosphamide, doxorubicin) +2xR (rituximab). Patients with ≥ 2 risk factors for CNS relapse or with occult meningeal involvement will be randomized in 1:1 ratio either into arm A with 2 cycles of prophylactic methotrexate 3g/m2 i.v., or into arm B with prophylactic 6x intrathecal methotrexate 12mg (1x intrathecal methotrexate in each cycle of systemic chemotherapy). Patients with 0-1 risk factor will be allocated into arm C without CNS prophylaxis. Patients will be observed for CNS relapse during the follow-up of 1year after the end of the first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed DLBCL
* age 18-72 years
* signed informed consent with the study
* first-line treatment 6 cycles of R CHOP +2x R or 6 cycles of DA EPOCH R+ 2xR

Exclusion Criteria:

* DLBCL and concomitant initial CNS involvement
* PMBL (primary mediastinal B-cell lymphoma)
* treatment with another chemotherapy than R CHOP or DA EPOCH R
* HIV positive, or active hepatitis B or C
* other concomitant serious disease (based on the decision of the physician-investigator)
* non-compliance of a patient
* any contraindication for application of anthracycline based chemotherapy or high dose methotrexate
* pregnancy or breast-feeding

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of CNS relapse in patients treated either with methotrexate i.v. or methotrexate i.t. or without CNS prophylaxis | 1 year

SECONDARY OUTCOMES:
Complete remission rate | 1 year
Overall response rate | 1 year
Overall survival | 2 years
Progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Mocikova, M.D., Ph.D., Principal Investigator — University Hospital Kralovske Vinohrady, Prague, Czech Republic; Marek Trněný, prof.M.D., Study Director — General University Hospital, Prague
Locations (6):
- Czechia (6):
  - University Hospital Brno-Bohunice, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - University Hospital Pilsen, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - General University Hospital Prague, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official Site of the Czech Lymphoma Study Group — http://www.lymphoma.cz
- Available data/document: Study Protocol — http://www.lymphoma.cz/docs/studies/dlbcl/CLSG-CNS-01_en.pdf